CLINICAL TRIAL: NCT07364799
Title: Effectiveness of the SoundHeal (Heal) Multi-Sensory Integrative Therapy in Enhancing Emotional Regulation Among Justice-Involved Youth and Its Effect on Therapeutic Alliance and Mental Health Outcomes
Brief Title: Effectiveness of the SoundHeal Multi-Sensory Integrative Therapy Among Justice-Involved Youth
Acronym: HEAL-SLOJSC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SoundHeal (Industry)
Collaborators: County of San Luis Obispo - Probation Department (Unknown); County of San Luis Obispo Health Agency (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHSLOSJC001
Record Dates: First submitted 2025-12-21; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Emotional Dysregulation; Therapeutic Alliance; Depression Disorder; Anxiety Disorders; Stress Disorders; Substance Use Disorders; Mental Health Disorders
Keywords: Emotional regulation; Emotional dysregulation; Justice-involved youth; Juvenile detention; Sensory-based intervention; multi-sensory stimulation therapy; Multisensory therapy; Sound therapy; music therapy; Vibroacoustic therapy; Therapeutic alliance; Therapy readiness; Mental health outcomes; substance use disorder; Coping skills; Non-verbal intervention; Journaling; Expressive Writing; Mindfulness
MeSH Terms: conditions — Anxiety Disorders; Stress Disorders, Traumatic; Substance-Related Disorders; Emotional Regulation | interventions — Wound Healing

STUDY DESIGN:
Intervention Model Description: This is a single-arm, open-label, pre-post study in which all enrolled participants receive the Heal intervention in addition to standard care, and outcomes are assessed by comparing within-participant changes from baseline to post-intervention over eight weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Heal Intervention (Experimental): Participants assigned to this arm will receive the Heal intervention in addition to standard care provided at the juvenile detention facility. The Heal intervention consists of brief, non-verbal, multi-sensory sessions delivered in a single-person booth (the Healpod), combining sound, music, gentle vibration, ambient light, and immediate expressive journaling or drawing prior to scheduled counseling sessions. All participants receive the intervention one to two times per week for approximately eight weeks, and outcomes are assessed using pre- and post-intervention measures.
  Interventions: Behavioral: Multi-sensory emotional regulation intervention (Heal)

INTERVENTIONS:
Behavioral: Multi-sensory emotional regulation intervention (Heal) — The multi-sensory emotional regulation intervention (Heal) is a brief, non-verbal behavioral intervention delivered in a single-person, distraction-free booth before scheduled counseling sessions. Each session includes approximately five minutes of calming sound and music, optional low-intensity vibroacoustic stimulation, and soft ambient lighting to support emotional regulation without requiring verbal processing or physical interaction with anyone.
  Immediately after each session, participants complete a brief writing activity (journaling or drawing) to reflect on their emotional state before, during and after the session. This reflective activity is used to support discussion during a standard therapy session with the clinician after.
  Sessions are delivered 1 to 2 times per week over eight weeks in addition to standard care. The intervention is non-invasive, supervised for safety, and may be stopped at any time. No medications or invasive procedures are involved.
  Other Names: Heal Intervention; Healpod intervention; Soundheal Intervention; Sensory-based emotional regulation intervention

SUMMARY:
Emotional dysregulation in justice-involved youth (JIY) is a condition that significantly impacts young people, their families, and juvenile justice and public health systems. Affecting an estimated 60-70% of detained Attention deficit hyperactivity disorderadolescents, it is a major driver of aggression, substance use, school failure, and later recidivism. Despite available treatments, managing emotional dysregulation in custody remains challenging, with youth often enduring high arousal, anger, and anxiety that persist into adulthood. Current popular therapies, including Cognitive Behavioral Therapy (CBT) and Dialectic Behavioral Therapy (DBT), often fall short in detention because they rely on verbal processing, require multiple scheduled sessions, and/or need highly trained staff. Other technologies, like biofeedback and neurostimulation techniques, are still under scrutiny for adolescents, given their higher-than-usual Adverse Events (AEs).

This SoundHeal study aims to evaluate a sensory intervention using the Healpod, a distraction-free physical space where a participant sits, delivering sound, music, gentle vibrations, and ambient light. Following this is a brief expressive journaling exercise to compare any before, during and after experience changes from the sensory immersion.

This prospective, single-center cohort study hypothesizes that these sessions will improve juveniles' ability to emotionally regulate, improve therapeutic alliance, mental health outcomes and build coping skills that can potentially help in long-term mental health and substance abuse treatment in JIY and beyond.

DETAILED DESCRIPTION:
Justice Involved Youth (JIY) often have difficulty with emotional regulation (ER) given all they go through physically, mentally and emotionally. Emotional dysregulation (ED) shows up as difficulty in managing anger and/or impulsivity and reacting rather than calmly responding to challenging situations faced negatively impacting their life.

Research consistently shows that incarcerated populations have far higher rates of ED and mental health disorders than the general youth population. The reason this is important in the context of this study is that ER difficulties act as a contributor to aggression and aggressive behaviors. In nationally representative JIY data, ED is the norm rather than the exception. In the "Survey of Youth in Residential Placement," 68% of confined youth reported being "easily upset" and 61% said they "lost their temper easily or felt angry a lot," clear, item-level indicators of ED among detained youth. By contrast, community studies show much lower rates for comparable constructs: the National Comorbidity Survey-Adolescent Supplement estimates 5.3-7.8% lifetime (and 1.7-6.2% 12-month) prevalence for intermittent explosive disorder, while clinical reviews put severe irritability in community youth at roughly 0.1-5%, and epidemiologic summaries place impairing emotional outbursts in about 4-10% of children and adolescents.

ED shows up as mental health disorders: a large meta-analysis of detained adolescents found strikingly elevated psychiatric morbidity with major depression (10.1% males, 25.8% females), Attention Deficit Hyperactivity Disorder (ADHD)(17.3% males, 17.5% females), and conduct disorder (~62% males, 59% females). By contrast, general U.S. youth have far lower trauma-related burden; for example, lifetime Post Traumatic Stress Disorder (PTSD) is about 5% overall (2.3% males, 8.0% females).

A very similar disproportion also shows up with substance use disorder (SUD) and alcohol use. According to a 2021 Substance Abuse and Mental Health Services Administration (SAMHSA) report, 7.5% of adolescents ages 12-17 had a SUD, 7% drank alcohol in the past month, and 14.1% adolescents drank alcohol in the past year. While this SAMHSA report did not have data on JIY, another 2023 report by the Bureau of Justice Statistics on drug and alcohol use stated that about 60% of youth met the criteria for SUD and 36% for alcohol use disorder, and that more than 63% met the criteria for severe SUD from 2008 to 2018.

Taken together, the data show that ED is not a side issue for JIY, it's a central, measurable driver of what derails treatment and destabilizes custody, conflict, impulsive reactions, misconduct, and worsening symptoms. Hence, there is a need for more effective innovative rehabilitation approaches that may help JIY strengthen ER, encourage therapeutic alliance, help improve mental health outcomes, develop healthy coping skills, and thereby potentially reduce recidivism and relapse rates in the long run.

SoundHeal's sensory-first intervention combines sound, music, gentle vibrations, and ambient light into a focused five-minute HealPod experience that helps bridge emotional dysregulation with mental-health and substance-use treatment.

The findings from this study aim to show that this structured approach can provide meaningful ER, improve therapeutic alliance, overcome mental health ailments, unlock engagement, and strengthen coping for youth who may otherwise remain resistant or disengaged in treatment.

The proposed study is intended to be an 8-week clinical trial. Participating juveniles will be selected from a single-site at SLO County Juvenile Hall for 12- to 18-year-old youth who are under residential treatment. Youth in this facility are ordered to stay 6-12 months and to receive intensive case management, treatment and educational services, making it the ideal population to work with within Juvenile Hall. Participating juveniles will be scheduled to use the Healpod 1-2 times a week before they meet their therapist. They will arrive 10 minutes before their scheduled session with their therapist, use the Healpod for about 5 minutes, and then journal/ write or draw about how they felt before, during and after the session. Therapists see the youth after their session and use the Heal journal as a starting point for talk therapy (Cognitive Behavioral Therapy/Dialectic Behavioral Therapy) treatment.

The Healpod (the tool for treatment) itself is a physical, rounded 4ft x 6ft telephone booth-like space equipped with speakers, low-frequency vibroacoustics, and a touchpad user interface for session selection. Once seated inside the Healpod, participants draw the curtains close and start their session.

The primary objective of this study is to measure ER and the secondary objectives to measure therapeutic engagement and mental health outcomes in treatment. While all show disparities between JIY and the general youth population, as discussed earlier, there is a cause-and-effect relationship between ER and engagement in treatment. The weight of evidence supports a directional, partly causal chain in which improving ER enables more engagement and adaptive coping, which then improves downstream outcomes.

Youth will fill out standardized questionnaires after their time inside the Healpod at the start, weekly, and at the end of the 8-week study period. Additionally, the therapist will fill out their assessment after talk therapy after their session with the youth.

ELIGIBILITY:
Inclusion Criteria:

* Age: Youth 12-18 years old. All participants enrolled in this study will be under the age of 18 at time of enrollment.
* Custody: Detained in SLO County, CA Juvenile Hall with at least 8 weeks of expected stay at the time the clinical trial starts
* Diagnosis: Documented history of being at risk or of having a history or current diagnosis of a mental health disorder (depression, anxiety, stress) and/or SUD
* Language/Comprehension: Basic English understanding; accommodations for limited literacy allowed
* Consent/Assent: Eligible juveniles must provide assent, with parent/guardian or Legally Authorized Representative (LAR) consent.
* Ensure that the person providing informed consent understands the information provided, even if that person providing informed consent agrees to be in the research.
* Participation: Willingness to comply with the Heal intervention, journaling, and questionnaires
* Recruitment and selection participation: Eligible participants will be selected in collaboration with facility behavioral-health staff using objective inclusion criteria only. Recruitment procedures are designed to be fair and free from arbitrary influence by facility administrators or peers.

Special Considerations: Because participants are minors and incarcerated, safeguards ensure voluntary participation, protection from coercion, age-appropriate communication, and accommodations for literacy or comprehension limits.

Exclusion Criteria:

* Age/Status: Not between 12-18 years old, or not currently detained in SLO County Juvenile Hall
* Length of Stay: Expected detention is less than 8 weeks at start of clinical trial
* Clinical Stability: Determined by onsite staff to be medically or psychiatrically unable to participate safely
* Consent/Assent: Unable to provide assent, or if parent/guardian or LAR does not provide consent
* If the person providing informed consent needs more time than is allowed by the research design.
* Language/Comprehension: Cannot understand basic English, even with literacy accommodations
* Participation: Unwilling to comply with the Heal intervention, journaling, or questionnaires
* Research staff will not personally use the device for research purposes. Their role is limited to facilitating device use for participants and monitoring protocol adherence.
* While the Healpod may be available for non-research use in other settings, this protocol strictly limits its use to the described research procedures. Any non-research use will be separated from this study, and no data will be collected from individuals outside of the study.
* Currently pregnant or becomes pregnant during the study period: If pregnant or pregnancy is discovered during participation, the individual will be withdrawn from the study to prevent any potential discomfort or unknown risk exposure related to the device environment (sound, vibration, or lighting).

Special Exclusions

* Juveniles whose participation may be influenced by coercion (e.g., enrollment tied to privileges or probation decisions)
* Juveniles with severe cognitive or behavioral impairment that prevents safe or meaningful participation

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change in Emotional Regulation | Baseline, midpoint (week 4 ±1), and end of intervention (week 8 or end of participation)
  Change in emotional regulation will be assessed using the Difficulties in Emotion Regulation Scale - 16 Item Version (DERS-16), a validated self-report questionnaire measuring difficulties in emotional awareness, clarity, impulse control, and access to emotion regulation strategies. Total scores range from 16 to 80, with higher scores indicating greater emotional dysregulation (worse outcome). The primary endpoint is change in DERS-16 total score from baseline to end of intervention.

SECONDARY OUTCOMES:
Change in Therapeutic Alliance | Baseline, midpoint (week 4 ±1), and end of intervention (week 8 or end of participation)
  Change in therapeutic alliance will be assessed using the Therapeutic Alliance Scale for Children - Revised (TASC-R), a validated youth-reported measure of perceived trust, collaboration, and engagement with the therapist. Total scores range from 12 to 48, with higher scores indicating a stronger therapeutic alliance (better outcome).
Change in Coping Skills | Baseline, midpoint (week 4 ±1), and end of intervention (week 8 or end of participation)
  Change in coping strategies will be assessed using the Kidcope Checklist of Coping Strategies (KidCOPE), a validated youth self-report measure of adaptive and maladaptive coping responses to stress. The scale includes multiple items rated for use of specific coping strategies, with total scores ranging from 0 to 30, with higher scores indicating greater use of coping strategies (better outcome).
Change in Depression Symptoms | Baseline and every two weeks during the intervention period (weeks 2, 4, 6, and 8)
  Change in depressive symptoms will be assessed using the Patient Health Questionnaire-9 (PHQ-9), a validated self-report measure of depressive symptom severity over the prior two weeks. Total scores range from 0 to 27, with higher scores indicating greater depressive symptom severity (worse outcome).
Change in Anxiety Symptoms | Baseline and every two weeks during the intervention period (weeks 2, 4, 6, and 8)
  Change in anxiety symptoms will be assessed using the Generalized Anxiety Disorder-7 (GAD-7), a validated self-report measure of anxiety severity. Total scores range from 0 to 21, with higher scores indicating greater anxiety symptom severity (worse outcome).
Change in Stress Symptoms | Baseline and every two weeks during the intervention period (weeks 2, 4, 6, and 8)
  Change in perceived stress will be assessed using the Perceived Stress Scale - 4 Item Version (PSS-4), a validated self-report measure of the degree to which situations in one's life are appraised as stressful. Total scores range from 0 to 16, with higher scores indicating greater perceived stress (worse outcome).
Change in Interoceptive Awareness | Baseline, midpoint (week 4 ±1), and end of intervention (week 8 or end of participation)
  Interoceptive awareness will be assessed using the Multidimensional Assessment of Interoceptive Awareness - Youth Version (MAIA-Y), a validated self-report measure assessing awareness of internal bodily sensations and their relationship to emotional and regulatory processes. Scale scores range from 1 to 6, with higher scores indicating greater interoceptive awareness and self-regulation (better outcome).

OTHER OUTCOMES:
Feasibility and Acceptability | Throughout the intervention period (up to 8 weeks)
  Feasibility and acceptability will be assessed through intervention adherence (number of sessions completed), therapist observations of engagement, and qualitative analysis of de-identified participant session journals.
Adverse Events (AEs) and Serious Adverse Events (SAEs) | Throughout the intervention period (up to 8 weeks)
  Safety will be assessed by monitoring and recording the number and type of adverse events and serious adverse events occurring during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Nishat Bhuiyan, PhD, Principal Investigator
Locations (1):
- San Luis Obispo County Juvenile Hall, San Luis Obispo, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sedlak, A. J., & McPherson, K. S. (2010). Youth's needs and services: Findings from the Survey of Youth in Residential Placement. Juvenile Justice Bulletin, Office of Juvenile Justice and Delinquency Prevention. https://www.ojp.gov/pdffiles1/ojjdp/227728.pdf
- [Background] Skinner-Osei, P., Mangan, L., Liggett, M., Kerrigan, M., & Levenson, J. S. (2019). Justice-involved youth and trauma-informed interventions. Justice Policy Journal, 16(2), 1-25. https://www.cjcj.org/media/import/documents/justice-involved_youth_and_trauma-informed_interventions.pdf
- [Background] Kelly EL, Novaco RW, Cauffman E. Anger and depression among incarcerated male youth: Predictors of violent and nonviolent offending during adjustment to incarceration. J Consult Clin Psychol. 2019 Aug;87(8):693-705. doi: 10.1037/ccp0000420. Epub 2019 Jun 17. PMID 31204840
- [Background] McLaughlin KA, Green JG, Hwang I, Sampson NA, Zaslavsky AM, Kessler RC. Intermittent explosive disorder in the National Comorbidity Survey Replication Adolescent Supplement. Arch Gen Psychiatry. 2012 Nov;69(11):1131-9. doi: 10.1001/archgenpsychiatry.2012.592. PMID 22752056
- [Background] Schreiber LR, Grant JE, Odlaug BL. Emotion regulation and impulsivity in young adults. J Psychiatr Res. 2012 May;46(5):651-8. doi: 10.1016/j.jpsychires.2012.02.005. Epub 2012 Mar 3. PMID 22385661
- [Background] Paulus FW, Ohmann S, Mohler E, Plener P, Popow C. Emotional Dysregulation in Children and Adolescents With Psychiatric Disorders. A Narrative Review. Front Psychiatry. 2021 Oct 25;12:628252. doi: 10.3389/fpsyt.2021.628252. eCollection 2021. PMID 34759846
- [Background] Saskovets M, Saponkova I, Liang Z. Effects of Sound Interventions on the Mental Stress Response in Adults: Scoping Review. JMIR Ment Health. 2025 Mar 24;12:e69120. doi: 10.2196/69120. PMID 40127440
- [Background] Dowdy R, Estes J, McCarthy C, Onders J, Onders M, Suttner A. The Influence of Occupational Therapy on Self-Regulation in Juvenile Offenders. J Child Adolesc Trauma. 2022 Nov 2;16(2):221-232. doi: 10.1007/s40653-022-00493-y. eCollection 2023 Jun. PMID 36340267
- [Background] Xiao X, Chen W, Zhang X. The effect and mechanisms of music therapy on the autonomic nervous system and brain networks of patients of minimal conscious states: a randomized controlled trial. Front Neurosci. 2023 May 12;17:1182181. doi: 10.3389/fnins.2023.1182181. eCollection 2023. PMID 37250411
- [Background] Rodriguez M, Kross E. Sensory emotion regulation. Trends Cogn Sci. 2023 Apr;27(4):379-390. doi: 10.1016/j.tics.2023.01.008. Epub 2023 Feb 15. PMID 36805103
- [Background] Krishnan C, Santos L, Peterson MD, Ehinger M. Safety of noninvasive brain stimulation in children and adolescents. Brain Stimul. 2015 Jan-Feb;8(1):76-87. doi: 10.1016/j.brs.2014.10.012. Epub 2014 Oct 28. PMID 25499471
- [Background] Caulfield, L.S. & Wilson, D. (2010). Female offenders' experiences of the arts in criminal justice. Journal of Social Criminology, 3, 67-90.
- [Background] Jennie L. Shufelt, M.S.; Joseph J. Cocozza, Ph.D. Youth with Mental Health Disorders in the Juvenile Justice System: Results From a Multi-State Prevalence Study.
- [Background] Daros AR, Haefner SA, Asadi S, Kazi S, Rodak T, Quilty LC. A meta-analysis of emotional regulation outcomes in psychological interventions for youth with depression and anxiety. Nat Hum Behav. 2021 Oct;5(10):1443-1457. doi: 10.1038/s41562-021-01191-9. Epub 2021 Sep 20. PMID 34545236
- [Background] Berking M, Ebert D, Cuijpers P, Hofmann SG. Emotion regulation skills training enhances the efficacy of inpatient cognitive behavioral therapy for major depressive disorder: a randomized controlled trial. Psychother Psychosom. 2013;82(4):234-45. doi: 10.1159/000348448. Epub 2013 May 22. PMID 23712210
- [Background] Compas BE, Jaser SS, Bettis AH, Watson KH, Gruhn MA, Dunbar JP, Williams E, Thigpen JC. Coping, emotion regulation, and psychopathology in childhood and adolescence: A meta-analysis and narrative review. Psychol Bull. 2017 Sep;143(9):939-991. doi: 10.1037/bul0000110. Epub 2017 Jun 15. PMID 28616996
- [Background] Shantakumari N, Ahmed M. Whole body vibration therapy and cognitive functions: a systematic review. AIMS Neurosci. 2023 May 18;10(2):130-143. doi: 10.3934/Neuroscience.2023010. eCollection 2023. PMID 37426779
- [Background] Eastburn, C. (2003). Gongs behind bars: Evaluation report of the Good Vibrations Gamelan in Prisons pilot project 2003. Wellingore: The Firebird Trust.
- [Background] Digard, L., Grafin von Sponeck, A. & Liebling, A. (2007). All Together Now: The therapeutic potential of a prison-based music programme. The Prison Service Journal, Issue 170, 3-14.
- [Background] Braun, V. & Clarke, V. (2006). Using thematic analysis in psychology. Qualitative Research in Psychology, 3, 77-101
- [Background] Chloe A. Greenbaum, Shabnam Javdani, Expressive writing intervention promotes resilience among juvenile justice-involved youth, Children and Youth Services Review, Volume 73, 2017, Pages 220-229, ISSN 0190-7409, https://doi.org/10.1016/j.childyouth.2016.11.034
- [Background] Chong HJ, Yun J. Music Therapy for Delinquency Involved Juveniles Through Tripartite Collaboration: A Mixed Method Study. Front Psychol. 2020 Oct 23;11:589431. doi: 10.3389/fpsyg.2020.589431. eCollection 2020. PMID 33192927
- [Background] Bryan K, Freer J, Furlong C. Language and communication difficulties in juvenile offenders. Int J Lang Commun Disord. 2007 Sep-Oct;42(5):505-20. doi: 10.1080/13682820601053977. PMID 17729143
- [Background] Allen CH, Kluger BM, Buard I. Safety of Transcranial Magnetic Stimulation in Children: A Systematic Review of the Literature. Pediatr Neurol. 2017 Mar;68:3-17. doi: 10.1016/j.pediatrneurol.2016.12.009. Epub 2017 Jan 4. PMID 28216033
- [Background] Fox, A. M., Miksicek, D., and Veele, S. (2019). An evaluation of Dialectical Behavior Therapy in Washington State's Juvenile Rehabilitation. Olympia, WA: Department of Children, Youth, and Families, Office of Innovation, Alignment, and Accountability.
- [Background] Folk JB, Yang P, Thomas A, Lyon J, Patel J, Yoon C, Barbara-Robles-Ramamurthy. Comprehensive Dialectical Behavior Therapy for Adolescents in a Juvenile Correctional Treatment Center: A Pilot Evaluation. Front Child Adolesc Psychiatry. 2023;2:1207575. doi: 10.3389/frcha.2023.1207575. Epub 2023 Nov 2. PMID 39220324
- [Background] Wadsworth ME. Development of Maladaptive Coping: A Functional Adaptation to Chronic, Uncontrollable Stress. Child Dev Perspect. 2015 Jun 1;9(2):96-100. doi: 10.1111/cdep.12112. PMID 26019717
- [Background] Michael B. Field, BJS Statistician; Elizabeth Davis, BJS Statistician; Amy D. Lauger, BJS Statistician Date Published July 2023 NCJ Number 305814
- [Background] Jamie R. Yoder; Kelly Whitaker; Camille R. Quinn. Perceptions of Recidivism Among Incarcerated Youth: The Relationship Between Exposure to Childhood Trauma, Mental Health Status, and the Protective Effect of Mental Health Services in Juvenile Justice Settings. Vol. 18 No. 1 (Spring 2017), 250-269, DOI: 10.18060/21305
- [Background] Okuda M, Picazo J, Olfson M, Hasin DS, Liu SM, Bernardi S, Blanco C. Prevalence and correlates of anger in the community: results from a national survey. CNS Spectr. 2015 Apr;20(2):130-9. doi: 10.1017/S1092852914000182. PMID 25831968
- [Background] Skinner-Osei et al. Justice Policy Journal, Fall, 2019 Justice-Involved Youth and Trauma-Informed Interventions. Justice Policy Journal. Volume 16, Number 2 (Fall, 2019) © Center on Juvenile and Criminal Justice 2019
- [Background] Melissa A. Brotman, Ph.D. brotman@mail.nih.gov, Katharina Kircanski, Ph.D., Argyris Stringaris, M.D., Ph.D., Daniel S. Pine, M.D., and Ellen Leibenluft, M.D. Publication: American Journal of Psychiatry Volume 174, Number 6 https://doi.org/10.1176/appi.ajp.2016.1607083
- [Background] Carlo Garofalo, Patrizia Velotti, Negative emotionality and aggression in violent offenders: The moderating role of emotion dysregulation, Journal of Criminal Justice, Volume 51, 2017, Pages 9-16, ISSN 0047-2352, https://doi.org/10.1016/j.jcrimjus.2017.05.015.
- [Background] Teplin LA, Abram KM, McClelland GM, Dulcan MK, Mericle AA. Psychiatric disorders in youth in juvenile detention. Arch Gen Psychiatry. 2002 Dec;59(12):1133-43. doi: 10.1001/archpsyc.59.12.1133. PMID 12470130
- [Background] Farnia, V., Golshani, S., Alikhani, M., & Akhondzadeh, S. (2023). Are there any possible side effects of neurofeedback? A systematic literature review and meta-analysis. Iranian Journal of Psychiatry and Behavioral Sciences, 17(4), e138064. https://doi.org/10.5812/ijpbs.138064
- [Background] Rahmani E, Rahmanian M, Mansouri K, Mokhayeri Y, Jamalpour Y, et al. Are There any Possible Side Effects of Neurofeedback? A Systematic Literature Review and Meta-analysis.Iran J Psychiatry Behav Sci.2023;17(3):e138064.https://doi.org/10.5812/ijpbs-138064.
- [Background] Duchschere JE, Reznik SJ, Shanholtz CE, O'Hara KL, Gerson N, Beck CJ, Lawrence E. Addressing a Mental Health Intervention Gap in Juvenile Detention: A Pilot Study. Evid Based Pract Child Adolesc Ment Health. 2023;8(2):236-251. doi: 10.1080/23794925.2022.2042873. Epub 2022 Apr 20. PMID 37637190
- [Background] Beaudry G, Yu R, Langstrom N, Fazel S. An Updated Systematic Review and Meta-regression Analysis: Mental Disorders Among Adolescents in Juvenile Detention and Correctional Facilities. J Am Acad Child Adolesc Psychiatry. 2021 Jan;60(1):46-60. doi: 10.1016/j.jaac.2020.01.015. Epub 2020 Feb 5. PMID 32035113

DOCUMENTS (2):
  • Study Protocol (2025-11-26): https://cdn.clinicaltrials.gov/large-docs/99/NCT07364799/Prot_000.pdf
  • Informed Consent Form (2025-12-02): https://cdn.clinicaltrials.gov/large-docs/99/NCT07364799/ICF_001.pdf